CLINICAL TRIAL: NCT01850693
Title: Prevalence and Characteristics of Coronary Atherosclerosis in Stroke Patients Using Coronary CT Angiography
Brief Title: Assessment of Coronary Artery Disease in Stroke Patients
Acronym: ACADIS
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Sponsor
Other Study IDs: NRF 2010-0023504
Record Dates: First submitted 2013-05-03; First posted 2013-05-09 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2013-05

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; stroke; coronary CT angiography
MeSH Terms: conditions — Coronary Artery Disease; Stroke

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Coronary artery disease, Stroke: Coronary artery disease, stroke, coronary CT angiography

SUMMARY:
This study is to evaluate the prevalence, plaque characteristics (plaque types, stenosis degree, remodeling) and predictors of coronary atherosclerosis in stroke patients with coronary CT angiography.

DETAILED DESCRIPTION:
Stroke and coronary artery disease (CAD) share common risk factors and pathological mechanisms. CAD is an important cause of death in patients with stroke.

Currently, coronary CT angiography (CCTA) is very useful non-invasive tool for detection of CAD and plaque analysis.

Therefore, the investigators aimed to evaluate the prevalence, plaque characteristics (plaque types, stenosis degree, remodeling) and predictors of CAD in stroke patients through follow-up (more than 5 years) using CCTA.

ELIGIBILITY:
Inclusion Criteria:

* Acute stroke patients who diagnosed by clinical and brain MR imaging
* Who performed coronary CT angiography within 3 months after acute stroke

Exclusion Criteria:

* intracranial hemorrhage including intracerebral, subdural or subarachnoid hemorrhage
* brain tumor
* Previous myocardial infarction
* Previously performed percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG) or other cardiac surgery
* Insufficient medical record
* Poor image quality of CCTA scan

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients on the basis of TOAST classification
Sampling Method: Non-Probability Sample
Enrollment: 1657 (Actual)
Dates: Start 2006-07; Primary Completion 2012-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
MACE (Major Adverse Cardiac Event) | Participants will be followed until June. 2015, an expeded average of 5 years
  MACE was included as follows: 1) all-cause mortality, 2) myocardial infarction, 3) unstable angina requiring hospitalization

SECONDARY OUTCOMES:
Any cardiac events | Participants will be followed until June. 2015, an expeded average of 5 years
  1) late revascularization: who underwent revascularization therapy mroe than 90days after CCTA and referral due ot new symptoms or an abnormal function test, 2) heart failure required hospitalization.

OTHER OUTCOMES:
Repeated stroke | Participants will be followed until June. 2015, an expeded average of 5 years
  newly developed stroke after CCTA scan

CONTACTS AND LOCATIONS:
Overall Officials: Eun Ju Chun, MD, Principal Investigator — Department of Radiology, Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea